CLINICAL TRIAL: NCT05412186
Title: Assessment of Reliability and Validity of Urdu Version of Cumberland Ankle Instability Tool Among Pakistani Patients Complaining for Ankle Sprain
Brief Title: Urdu Version Of Cumberland Ankle Instability Tool: Reliability And Validity Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00277
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Ankle Sprains
Keywords: Cumberland Ankle Instability Tool; Urdu Version; Reliability; Validity; Ankle Sprains; Ankle Instability
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to check reliability and validity, of translated Urdu version of the Cumberland Ankle Instability Tool develop and test its psychometric properties and responsiveness in Urdu speaking population in Pakistan endure with Ankle sprain and ankle instability complaints.

DETAILED DESCRIPTION:
The Urdu version of the Cumberland Ankle Instability Tool will be translated and dignified for internal reliability test-retest consistency and cross cultural guidelines of self-reported measures, to evaluate validity (convergent and discrimination)of the sample of 125 participants who experience ankle sprain, participants choose by convenience sampling technique reinforced on already elaborated inclusion/exclusion criteria.Evaluation Form will be filled by a patient twice an day by observer for inter observer assessment , with an interval of 30 minutes to 2 hours between the first and second application. Third assessment will be carried out after 7 days obtained by 1st Observer (re-testing),they completed Cumberland Ankle Instability Tool Urdu version who had ankle sprain in past 3 months and also its correlation checked with lower extremity functional scale, visual analogue scale, and Short Form - 36 short form health survey participant also completed these scales, In general population with ankle sprain and ankle instability in this study we intended to translate the original version of Cumberland Ankle Instability Tool into Urdu cross- culturally adaptation and examine psychometric properties and cut-off score of the Cumberland Ankle Instability Tool Urdu version.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are 18 years of age and
* Participants who were able to understand and complete the self-reported questionnaires (native Urdu speakers, with at least 8 years of education).

Exclusion Criteria:

* People who have ankle sprain episode and/or lower extremity injury within the last 2 months and/or any neurological or neuromuscular disease.
* Participants were also excluded if they did not fill out 2 or more questions of the Urdu Version Of Cumberland Ankle Instability Tool

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study subjects of this research will be the general population of having ankle sprain.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-08-10 (Estimated); Study Completion 2022-08-12 (Estimated)

PRIMARY OUTCOMES:
Cumberland Ankle Instability Tool | 1st day
  The Cumberland Ankle Instability Tool is combined of 9 items with multiple options decrease patient obligation and increase reliability, related to different aspects of Cumberland Ankle Instability such as ankle pain, daily sports physical activities may cause Ankle sprain, subjective instability, and the response of the ankle to episodes of generous means.The instrument extent sum scores from 0 (severe instability) to 30 (ankle totally stable).
Lower Extremity Functional Scale | 1st day
  The lower extremity functional scale is a well-known and validated patient-rated outcome measure for measuring lower extremity function
Visual Analogue Scale | 1st day
  A Visual Analogue Scale is a measurement tool that attempts to quantify a feature or attitude that is thought to range throughout a continuum of values but is difficult to measure directly.
Short Form Health Survey - 36 | 1st day
  The Short form health survey is a 36-question multipurpose short-form health assessment. It produces an 8-scale score profile as well as summary metrics. It's a broad measure of health rather than one that focuses on a specific age, condition, or treatment group. It produces an eight-scale profile of scores as well as summary indicators of physical and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No